CLINICAL TRIAL: NCT00760019
Title: Inflammation and Vascular Function in Atherosclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua A. Beckman, MD, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005P-001406; NCT00762827 (obsolete NCT alias)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Atherosclerosis
Keywords: vascular inflammation; endothelium-dependent flow-mediated blood vessel function
MeSH Terms: conditions — Atherosclerosis | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salsalate first, then Placebo (Active Comparator): In this crossover study, this group was randomly allocated therapy with salsalate first, a 4 week washout, then 4 weeks of placebo therapy in a double-blinded fashion.
  Interventions: Drug: salsalate
- Placebo first, then Salsalate (Placebo Comparator): In this crossover study, this group was randomly allocated therapy with placebo first, a 4 week washout, then 4 weeks of salsalate therapy in a double-blinded fashion.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: salsalate — 1.5 grams orally 3 times daily
  Other Names: Disalcid
  Arms: Salsalate first, then Placebo
Drug: placebo — matching placebo
  Arms: Placebo first, then Salsalate

SUMMARY:
The purpose of this study is to determine whether reducing inflammation in blood vessels with an aspirin-like drug called salsalate will improve blood vessel function.

DETAILED DESCRIPTION:
To test the hypothesis that inhibition of I [kappa] B kinase [beta] (IĸKβ), an inflammatory mediator, by high dose salsalate, will restore insulin-mediated endothelium-dependent vasodilation in subjects with atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking adult subjects with known atherosclerosis

Exclusion Criteria:

* Uncontrolled hypertension (> 140/90 mmHg)
* Untreated hypercholesterolemia (LDL > 160 mg/dL)
* Diabetes mellitus
* Alanine Aminotransferase > 150
* Creatinine > 1.4 mg/dL
* Concommitant use of warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-08; Primary Completion 2009-10 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A. Beckman, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sullivan AE, Courvan MCS, Ada AW, Wasserman DH, Niswender KD, Shardelow EM, Wells EK, Wells QS, Freiberg MS, Beckman JA. The Role of Serum Free Fatty Acids in Endothelium-Dependent Microvascular Function. Endocrinol Diabetes Metab. 2025 Mar;8(2):e70031. doi: 10.1002/edm2.70031. PMID 39888728
- [Derived] Nohria A, Kinlay S, Buck JS, Redline W, Copeland-Halperin R, Kim S, Beckman JA. The effect of salsalate therapy on endothelial function in a broad range of subjects. J Am Heart Assoc. 2014 Jan 3;3(1):e000609. doi: 10.1161/JAHA.113.000609. PMID 24390146

RESULTS

PARTICIPANT FLOW:
Groups:
- Atherosclerosis/Metabolic Syndrome: Salsalate First, Then Plac: Subjects with either Metabolic Syndrome/Atherosclerosis received either 4.5 g/day salsalate for 4 weeks, washout for 4 weeks, and matching placebo for 4 weeks.
- Atherosclerosis/Metabolic Syndrome: Placebo First, Then Salsal: Subjects with either Metabolic Syndrome/Atherosclerosis received placebo for 4 weeks, washout for 4 weeks, and 4.5 g/day salsalate for 4 weeks.
- Healthy Subjects: Salsalate First, Then Placebo: Healthy subjects received either 4.5 g/day salsalate for 4 weeks, washout for 4 weeks, and matching placebo for 4 weeks.
- Healthy Subjects: Placebo First, Then Salsalate: Healthy subjects received placebo for 4 weeks, washout for 4 weeks, and 4.5 g/day salsalate for 4 weeks.
Period: Overall Study
Arm/Group | Atherosclerosis/Metabolic Syndrome: Salsalate First, Then Plac | Atherosclerosis/Metabolic Syndrome: Placebo First, Then Salsal | Healthy Subjects: Salsalate First, Then Placebo | Healthy Subjects: Placebo First, Then Salsalate
Started | 15 | 15 | 14 | 14
Completed | 15 | 15 | 14 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atherosclerosis or Metabolic Syndrome: Participant flow is identical to that of NCT00762827 ("The Impact of Reducing Inflammation on Vascular Function in the Metabolic Syndrome"):
  The study arms reflect the randomized, placebo-controlled, double-blinded crossover design of the study. In this arm, individuals with either Metabolic Syndrome or Atherosclerosis received either 4.5 g/day salsalate or matching placebo for a 4-week long period. After a 4-week washout interval, these individuals crossed over and received either the salsalate or the placebo (whichever they did not receive in the first study period) for another 4 weeks.
- Healthy: Participant flow is identical to that of NCT00762827 ("The Impact of Reducing Inflammation on Vascular Function in the Metabolic Syndrome"):
  The study arms reflect the randomized, placebo-controlled, double-blinded crossover design of the study. In this control arm, healthy individuals received either 4.5 g/day salsalate or matching placebo for a 4-week long period. After a 4-week washout interval, these individuals crossed over and received either the salsalate or the placebo (whichever they did not receive in the first study period) for another 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Atherosclerosis or Metabolic Syndrome | Healthy | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9) | 52 (13) | 56 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated, Endothelium-dependent Vasodilation
Description: Flow-mediated, endothelium-dependent vasodilation (percentage increase in brachial artery diameter after a 5 minute ischemic stimulus) measured at the end of placebo treatment and end of salsalate treatment were compared.
Time Frame: Upon completion of 4 weeks of salsalate and placebo treatment
Population: The ultrasound data for two subjects was inadequate for analysis. This determination was made prior to unblinding. The data for these two subjects were discarded, leaving 56 subjects for analysis.
Measure: Median (Inter-Quartile Range); unit: percentage vasodilation
Groups:
- Salsalate; Placebo: Outcomes were measured at the end of each 4-week study period. Here, median flow-mediated, endothelium-dependent vasodilation after 4 weeks of 4.5 g/day salsalate is compared with median FMD after 4 weeks of matching placebo. Data represent all subjects: those with atherosclerosis/metabolic syndrome as well as healthy controls.
Arm/Group | Salsalate | Placebo
Number analyzed (Participants) | 56 | 56
percentage vasodilation | 6.8 [5.2 to 12.0] | 8.7 [5.4 to 13.5]

ADVERSE EVENTS:
Groups:
- Salsalate: Adverse Event Data represent all subjects: those with atherosclerosis/metabolic syndrome as well as healthy controls that received Salsalate
- Placebo: Adverse Event Data represent all subjects: those with atherosclerosis/metabolic syndrome as well as healthy controls that received Placebo
Arm/Group | Salsalate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 6/58 | 0/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate (N=58) | Placebo (N=58)
Tinnitus (Ear and labyrinth disorders) | 6 (6) | 0 (0) — 6 participants had study drug dose reduced to 3 g/day due to tinnitus, which resolved after dose reduction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No